CLINICAL TRIAL: NCT06742944
Title: Draw-10: A Weekly Blood Draw Study to Understand the Biological Variability of Plasma pTau-217
Acronym: Draw-10
Status: Completed | Type: Observational
Sponsor: Banner Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: API-0002; R01AG058468 (NIH)
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
Keywords: plasma pTau217
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — frozen plasma blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants age 50-80 with normal cognition or mild impairment: All participants will provide 10 plasma samples over the course of 9 weeks. This is an observational cohort study (no intervention(s) administered)

SUMMARY:
This is an observational study that will serially collect 10 plasma samples over the course of 9 weeks from the same individuals to assess fluctuations in blood biomarker results.

DETAILED DESCRIPTION:
Blood biomarkers offer a less invasive and cheaper method for identifying Alzheimer's disease (AD)-related changes. Already, blood biomarkers for AD are being adopted by clinical practice and their use will only expand in coming years. However, blood biomarkers are susceptible to fluctuations not yet well characterized. Such fluctuations, although rarely observed in current research settings, may influence the biological evaluation of dementia once implemented into routine settings. The study at present aims to identify how blood biomarkers fluctuate over a short period of time in the same individual and assess drivers of these fluctuations.

ELIGIBILITY:
Inclusion Criteria:

* able and wiling to provide informed consent
* Aged 50-80 years old at the time of signing study consent; participants aged 50-59 years will be no more than 20% of the total study population
* Has normal cognition or mild impairment at screening MoCA by a score of greater than or equal to 18; participants with a Montreal Cognitive Assessment (MoCA Test) score between 18-25 will be no more than 20% of the total study population
* able and wiling to fully comply with study procedures defined in the protocol
* Written and spoken fluency in English

Exclusion Criteria:

* Plans to begin any new treatment or is having surgery during the 9-week draw timeframe
* Currently enrolled in a clinical trial using an investigational drug

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Arizona residents
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Fluctuations in plasma pTau217 biomarker results | 9 weeks
  Assess within participant changes in plasma pTau217 biomarker assay levels over the course of the study
Frequency of large unknown biomarkers spike | 9 weeks
  Determine the frequency of large, unknown biomarkers spike that would influence a clinical decision.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica B Langbaum, PhD, Principal Investigator — Banner Alzheimer's Institute
Locations (2):
- United States (2):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Alzheimer's Institute Tucson, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: Yes
study dataset and biological samples will be shared with qualified investigators
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared within 12 months after study completion